CLINICAL TRIAL: NCT02812901
Title: Morning / Afternoon Variation in Myocardial Ischemia Tolerance
Brief Title: Tolerance of Myocardium to Ischemia Injury
Acronym: TOMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-56; 2015-A00864-45 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-06-22; First posted 2016-06-24 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2017-08

CONDITIONS: Reperfusion Injury; Myocardial Ischemia
MeSH Terms: conditions — Reperfusion Injury; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- morning group (Other): cardiac surgery scheduled in the morning
  Interventions: Procedure: cardiac surgery scheduled in the morning
- afternoon group (Other): cardiac surgery scheduled in the afternoon
  Interventions: Procedure: cardiac surgery scheduled in the afternoon

INTERVENTIONS:
Procedure: cardiac surgery scheduled in the morning — cardiac surgery scheduled in the morning
  Arms: morning group
Procedure: cardiac surgery scheduled in the afternoon — cardiac surgery scheduled in the afternoon
  Arms: afternoon group

SUMMARY:
This study aims to understand the impact of time-of-the day on human myocardial tolerance to ischemia-reperfusion by exploring atrial myocardium biopsied during cardiac surgery. Patients scheduled for non-urgent cardiac surgery (coronary artery by-pas graft and/or aortic valve replacement) will be assigned to a morning or an afternoon cardiac surgery based on randomization. Myocardial biopsies will be explored in ex vivo conditions mimicking ischemia-reperfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for coronary artery bypass graft surgery and/or aortic valve replacement with extra-corporeal circulation
* Patient in sinus rhythm at the time of surgery
* Patient older than 18
* Patient able to understand the information and consent forms

Exclusion Criteria:

* Medical history of type 2 diabetes, atrial fibrillation or use of class III anti-arhythmic drug
* left ventricle ejection fraction < 40%
* Pregnancy
* Patient in emergency condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
ischemia reperfusion injury in ex vivo conditions | the day of the myocardial biopsy
  measurement of hs troponin T released by the myocardium samples in the superfusion solution after ex vivo conditions mimicking ischemia-reperfusion

CONTACTS AND LOCATIONS:
Overall Officials: David Montaigne, MD, PhD, Principal Investigator — Lille University Hospital
Locations (1):
- Lille University Hospital, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Montaigne D, Marechal X, Modine T, Coisne A, Mouton S, Fayad G, Ninni S, Klein C, Ortmans S, Seunes C, Potelle C, Berthier A, Gheeraert C, Piveteau C, Deprez R, Eeckhoute J, Duez H, Lacroix D, Deprez B, Jegou B, Koussa M, Edme JL, Lefebvre P, Staels B. Daytime variation of perioperative myocardial injury in cardiac surgery and its prevention by Rev-Erbalpha antagonism: a single-centre propensity-matched cohort study and a randomised study. Lancet. 2018 Jan 6;391(10115):59-69. doi: 10.1016/S0140-6736(17)32132-3. Epub 2017 Oct 26. PMID 29107324